CLINICAL TRIAL: NCT06971744
Title: Autophagy Maintenance (AUTOMAIN) Therapy in High-Grade Serous Ovarian Cancer: A Phase II Trial
Brief Title: Autophagy Maintenance (AUTOMAIN)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103919; Pro00143653 (Other: Medical University of South Carolina)
Record Dates: First submitted 2025-04-03; First posted 2025-05-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hydroxychloroquine; Nelfinavir; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hydroxychloroquine+Nelfinavir+Bevacizumab (Experimental): Subjects will take Hydroxychloroquine 3x 200 milligram tablets twice daily Subjects will take Nelfinavir 2x 625 milligram tablets twice daily Subjects will be administered Bevacizumab IV 15 milligram/kilogram every 3 weeks.
  DLT Period 21 Days (1 Cycle)
  Interventions: Drug: Hydroxychloroquine; Drug: Nelfinavir; Drug: Bevacizumab

INTERVENTIONS:
Drug: Hydroxychloroquine — 3 x 200 milligram tablets twice daily
Drug: Nelfinavir — 2x 625 milligram tablets twice daily
Drug: Bevacizumab — IV 15 milligram/kilogram every 3 weeks

SUMMARY:
This is a single-institution, single-arm study with a safety lead-in to determine if previously established safe doses of autophagy drugs, hydroxychloroquine (HCQ) and nelfinavir mesylate (NFV) will benefit ovarian cancer patients in a maintenance setting. Patients will receive the two study drugs HCQ and NFV in combination with maintenance bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have platinum-sensitive first recurrent high-grade serous or high-grade predominantly serous ovarian cancer, fallopian tube cancer, or primary peritoneal cancer. Patients must have had a 6-month disease-free progression since last platinum chemotherapy to be considered platinum sensitive.
* All participants must agree to have previously undergone genetic testing with germline panel testing with at least BRCA 1/2 mutation status known and/or somatic tumor next generation sequencing with homologous recombination deficiency (HRD) testing and/or loss of heterozygosity (LOH) known.
* Participants must be enrolled within 3-8 weeks of the first day of the last cycle of platinum-based chemotherapy for their first cancer recurrence. - Participants must have received at least 3-courses of bevacizumab during chemotherapy and have a plan to continue maintenance bevacizumab therapy.
* Evidence of platinum-sensitive response to current platinum-based chemotherapy with a partial or complete response based on imaging or CA-125 trend
* Participants of childbearing potential must have a negative serum or urine pregnancy test (beta human chorionic gonadotropin [hCG]) within 7 days before receiving the first dose of study treatment.
* Voluntary, signed, and dated, Institutional Review Board (IRB) approved consent form per regulatory and institutional guidelines.
* 18 years of age or older.
* ECOG performance status of 0-2
* Bilirubin ≤ 1.5 times the upper limit of normal (ULN) and AST / ALT ≤ 3 times ULN. Subjects with Gilbert's syndrome may be included if the total bilirubin is < 3 times ULN and the direct bilirubin is within normal limits.
* CrCl ≥35 mL/min, according to the Cockgroft-Gault formula.
* Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3.
* Platelet count ≥ 75,000 cells / mm3
* Hemoglobin ≥ 9 g/ dL, recent transfusion is allowed, though must be ≥ 7 days C1D1 of investigational agents
* Adequately controlled blood pressure (<160 mm Hg/100 mm Hg) as determined by the treating investigator.
* Subjects with the potential to produce children must agree to effective contraceptive method use during study participation and at least 6 months after discontinuation of the study.
* Patients requiring narcotic analgesics must be on stable doses for at least 2 weeks before study entry.
* Patients must discontinue any statin use within 48 hours of beginning study treatment.
* Patients must have a QT interval of <450 ms on screening upon ECG.
* Patients who have diabetes mellitus must have it well-controlled (A1c of <8%).

Exclusion Criteria:

* New York Heart Association (NYHA) Class III or IV cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or history of ischemia on baseline ECG.
* Underlying psychiatric disorder requiring hospitalization within the last two years.
* Clinically significant neurological disorder (Parkinson's disease, dementia, multiple sclerosis), as determined by the enrolling investigator.
* Platinum resistant or refractory disease
* Active, uncontrolled bacterial, viral, or fungal infection, requiring systemic therapy.
* Treatment with local or systemic radiation therapy, surgery, or investigational therapy within 28 days before registration with the exception of the platinum doublet and bevacizumab.
* Unwillingness or inability to comply with procedures required in this protocol.
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the Investigator.
* Patients who are receiving coumadin
* Patients who are currently participating in any other clinical trial of an investigational product.
* Any other mental incapacitation or psychiatric illness that would preclude study participation, as determined by the enrolling investigator.
* Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled in this study.
* Female patients who are of child-bearing potential (WOCBP) who are pregnant or planning to become pregnant during the study or within 6 months of the last dose of study drugs. A urine pregnancy test for WOCBP will be collected during the screening period. Females will be determined not to be of child-bearing potential with a history of hysterectomy, tubal ligation, dual salpingo-oophorectomy, or age 45 or older with postmenopausal status > 12 months.
* Patients unable to stop taking strong inhibitors and inducers of CYP2C8, CYP3A4, CYP2C19, CYP2D6, FMO-1, and MAO-A.
* Patients unable to stop taking substrates of CYP2D6, CYP3A4, P-gp, MATE1K, and MATE2K.
* Patients diagnosed with myasthenia gravis
* Patients with G6PD Deficiency
* Patients with porphyria
* Platinum-sensitive patients that are candidates for PARP inhibitor maintenance, patients will be allowed if previously did not tolerate PARP and opt against PARP maintenance
* Patients that have contraindications to bevacizumab, as per approved product labeling
* Patients that have a high ASCVD score based on the American College of Cardiology ASCVD Risk Estimator Plus calculator and who should not stop their statin due to cardiovascular risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-06-18 (Estimated); Study Completion 2029-06-18 (Estimated)

PRIMARY OUTCOMES:
Safety of combination of study drugs | 6 months
  To measure the safety of HCQ + NFV in combination with standard-of-care maintenance bevacizumab in patients with high-grade serous ovarian cancer. DLT (dose limiting toxicity) is the standard endpoint in evaluating safety at this study phase. Will monitor adverse events per CTCAE v5.0.
Evaluation of Anti Tumor Activity | 6 months
  Evaluate the anti-tumor activity of HCQ + NFV in combination with standard-of-care maintenance bevacizumab in patients with high-grade serous ovarian cancer. Measured by 6-month progression-free survival rate, a composite metric based on CA 125 and radiographic imaging.

SECONDARY OUTCOMES:
Changes in CA125 | 6 months
  changes in CA125 in patients treated with HCQ + NFV in combination with standard-of-care maintenance bevacizumab
Changes in Quality of Life | 6 months
  To document the change in QOL (via disease-specific FACT questionnaire, composite score) in patients treated with HCQ + NFV in combination with standard-of-care maintenance bevacizumab

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States